CLINICAL TRIAL: NCT03261362
Title: Branched-Chain Amino Acid Dietary Reduction Under Weight Maintainance in Overweight Patients With Type 2 Diabetes
Brief Title: Impact of Branched-chain Amino Acids in the Development of Insulin Resistance
Acronym: BRAAWO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Diabetes Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2014092783
Record Dates: First submitted 2017-08-22; First posted 2017-08-25 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Amino acid powder with all amino acids (Placebo Comparator): amino acid powder 80 g oral Administration 1 week
  Interventions: Dietary Supplement: Branched-chain amino acids reduced intake
- Amino acid powder without BCAAs-reduced intake (Active Comparator): Branched-chain amino acids reduced intake - amino acid powder lacking BCAAs 80 g oral Administration 1 week -
  Interventions: Dietary Supplement: Branched-chain amino acids reduced intake

INTERVENTIONS:
Dietary Supplement: Branched-chain amino acids reduced intake

SUMMARY:
The purpose of this study is to clarify the role of the branched-chain amino acids in the development of Insulin resistance in patients with diabetes

DETAILED DESCRIPTION:
The proposed project aims to elucidate the role of the BCAA in the development of insulin resistance and type 2 diabetes. The project tests the hypothesis that a diet induced decrease of BCAAs concentrations alter the metabolic mechanisms involved in the control insulin resistance and diabetes progression.

The specific aims are to elucidate the effect of the diet induced decrease of BCAAs concentrations on (I) peripheral and hepatic insulin sensitivity (II) ectopic fat distribution (III) energy metabolism (IV) metabolic and inflammatory status

ELIGIBILITY:
Inclusion Criteria:

* Diabetes type 2
* Non smokers
* Untrained
* Willingness to adhere to a diet intervention

Exclusion Criteria:

* Chronic disease
* Pregnancy
* Cancer
* Antibiotic therapy
* Drug/alcohol abuse
* Competitive athletes

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Clamp test | up to 24 weeks
  Insulin sensitivity test

SECONDARY OUTCOMES:
Mixed Meal Test | up to 24 weeks
  B cell function test

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, MD, Principal Investigator — Deutsches Diabetes Zentrum
Locations (1):
- German Diabetes Centre, Düsseldorf, Germany

REFERENCES:
- [Derived] Karusheva Y, Koessler T, Strassburger K, Markgraf D, Mastrototaro L, Jelenik T, Simon MC, Pesta D, Zaharia OP, Bodis K, Barenz F, Schmoll D, Wolkersdorfer M, Tura A, Pacini G, Burkart V, Mussig K, Szendroedi J, Roden M. Short-term dietary reduction of branched-chain amino acids reduces meal-induced insulin secretion and modifies microbiome composition in type 2 diabetes: a randomized controlled crossover trial. Am J Clin Nutr. 2019 Nov 1;110(5):1098-1107. doi: 10.1093/ajcn/nqz191. PMID 31667519